CLINICAL TRIAL: NCT04066686
Title: Evaluation on the Level of Discomfort and Restriction on Activities of Daily Living (ADLs) Whilst C-spine Immobilised in a Spinal Collar After C-spine Injury.
Brief Title: Evaluation of Comfort in a Spinal Collar
Status: Completed | Type: Observational
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18SM4650
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Results first posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Neck Injuries
Keywords: Neck Injuries
MeSH Terms: conditions — Neck Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young: Participants recruited into one of two groups on age stratification. Young cohort defined as aged 18-65yrs old
- Elderly: Participants recruited into one of two groups on age stratification. Elderly cohort defined as over 65yrs of age.

SUMMARY:
This is an observational study which aims to assess the comfort of a spinal collar in patients who have them fitted as part of their clinical care due to neck injury.

DETAILED DESCRIPTION:
The study follows the patient journey including long term follow up (up to 120 days following admission). The information gathered will be from the standard clinical care delivered and include demographics, baseline function, the injuries sustained following trauma and prescribed analgesia with records of the most recent time and dose administered. Any scans done of the neck for clinical purposes will be anonymised and analysed for measurements of angulation. In addition to this there will be a survey on the comfort of the collar and of their functional ability at the current time at various points during their inpatient admission.

ELIGIBILITY:
Inclusion Criteria:

1. All patients aged 18yrs and over with a C-spine injury immobilised in a spinal collar
2. Patients must be nursed on Major Trauma Ward
3. Ability to give informed consent to participate in the study.

Exclusion Criteria:

1. Patients under 18yrs age
2. Patients who lack capacity to consent for entry into the study
3. Patients who are receiving level 2( High dependency unit) or level 3 (Intensive care unit) clinical care
4. Patients who are unable to complete the visual analogue score or questionnaire due to having co-existent severe hearing and visual impairment. Severe hearing impairment will be defined as unable to hear the researcher with hearing aids if required. Severe visual impairment will be defined as being unable to read the patient information sheet even with visual aids.
5. Patients unable to understand the patient leaflet in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18yrs and over who are admitted to St Mary's Hospital with a C-spine injury will be invited to participate
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fertleman, Principal Investigator — Study Principal Investigator Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Heathcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Young | Elderly
Started | 14 | 13
Completed | 12 | 13
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participant withdrawal led to a reduction in the overall number of participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Young | Elderly | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 0 | 12
  >=65 years | 0 | 13 | 13
Age, Continuous [Median (Full Range); unit: years] | 47 [23 to 64] | 75 [65 to 90] | 65.5 [23 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 11 | 7 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Measurement of the Level of Discomfort Produced by the Spinal Collar in Adult Patients With a C-spine (Neck) Injury.
Description: 'Visual Analogue Scale' for pain (self reported: minimum 0=no pain at all, maximum 10= worst pain imaginable)
Time Frame: During inpatient admission (an average of two weeks)
Population: 11 Young participants and 9 Elderly participants completed the visual analogue score (some participants chose not to complete the score). Visual analogue score was assessed at single time point during the study.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Young | Elderly
Number analyzed (Participants) | 11 | 9
score on a scale | 1 [0 to 8] | 4.9 [0 to 9]

2. Secondary Outcome: Measurement of Change of Impedance on Activities of Daily Living Produced by the Spinal Collar in Adult Patient With a C-spine (Neck) Injury.
Description: 'Neck Disability Index' Questionnaire (Validated functional assessment which consists of ten questions to assess how that persons neck pain affects abilities in everyday life. It is a questionnaire format with multi-choice answer options). Minimum score = 0, Maximum score = 50. The overall percentage score is calculated as follows: e.g. 16 (total scored) divided by 50 (total possible score) x 100 = 32%. A higher percentage indicates a worse outcome i.e. higher disability.
Time Frame: At baseline (retrospectively) and at time of wearing the spinal collar after injury
Population: Only 10 participants in the Young group and 6 participants in the Elderly group were able to complete the 'Neck Disability Index' Questionnaires (retrospectively for baseline and at the time of wearing the spinal collar after injury).
Measure: Mean (Full Range); unit: percentage score on a scale
Arm/Group | Young | Elderly
Number analyzed (Participants) | 10 | 6
percentage score on a scale
  At baseline | 8.99 [0 to 30] | 6.28 [0 to 17.7]
  Wearing the spinal collar after injury | 50.83 [0 to 78] | 35.67 [4 to 62.5]

3. Secondary Outcome: Measurement of Spinal Angulation
Description: Measurements of angulation between specified bony anatomical landmarks to investigate degree of curvature within the C-spine performed on any neck imaging completed as part of routine clinical care. Statistical analysis to allow comparison of young and elderly groups.
Time Frame: Through study completion, up to one year
Population: Data not available
Arm/Group | Young | Elderly
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Duration of study - 7 months
Arm/Group | Young | Elderly
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT04066686/Prot_000.pdf